CLINICAL TRIAL: NCT05749809
Title: The Relationship Between Lower Extremity Selective Motor Control and Gait in Children With Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_05
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to examine the relationship between lower extremity selectivity and gait in children with cerebral palsy. 32 volunteer children with CP between the ages of 5-20 will participate in the study. The Selective Control Assessment of the Lower Extremity (SCALE) questionnaire will be used to assess lower extremity selectivity, and the Edinburgh observational gait scale will be used to assess gait. Both assessments are observational.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5-20
* Diagnosed with CP

Exclusion Criteria:

* Medical complications that limit participation in assessments (for example, severe visual impairment)
* Lower extremity surgery or botox surgery in the last 6 months
* Mental problems that cannot understand the commands given

Ages: 5 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Visual Gait Score | Baseline
  It consists of 17 items scored separately for the right and left lower extremities. Assessments include 6 anatomical levels: trunk, pelvis, hip, knee, ankle, and foot. These anatomical levels are evaluated in the sagittal, coronal and transverse planes. A 3-point ordinal scale is used for scoring. In scoring, a value of 0 indicates normal, a value of 1 indicates moderate deviation from normal, and a value of 2 indicates significant deviation from normal. The scores obtained by watching the camera recordings for each lower extremity are summed and a single score is obtained.
Selective Control Assessment of the Lower Extremity (SCALE) | Baseline
  Evaluates the selective motor control of the lower extremities. It evaluates hip, knee, ankle, subtalar and finger joints bilaterally. Voluntary flexion and extension movements are observed to assess selective voluntary motor control at each joint. Except for the hip joint, which is tested in the side-lying position to allow adequate joint movement, the evaluation of other joints is made in the sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)